CLINICAL TRIAL: NCT04173390
Title: Preemptive Analgesia With Pregabalin in Heart Surgery: a Randomized Clinical Trial
Brief Title: PREemptive Analgesia With preGABAlin in HEART Surgery
Acronym: PREGABA-HEART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Bruno Robalinho Cavalcanti Barbosa, Principal Investigator, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDC DT 023/19/122; 17907319.5.0000.8069 (Registry Identifier: PLATAFORMA BRASIL)
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pregabalin (Experimental)
  Interventions: Drug: Pregabalin 150mg
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Pregabalin 150mg — Preemptive use of pregabalin 150 mg starting three days before surgery up to the third postoperative day
  Arms: pregabalin
Drug: Placebo oral tablet — Preemptive use of Placebo oral tablet starting three days before surgery up to the third postoperative day
  Arms: placebo

SUMMARY:
BACKGROUND: Postoperative pain after cardiac surgery has high incidence and is associated with worse morbidity. Pregabalin is a new antiepileptic drug used in patients with chronic pain and has been studied even more in postoperative. OBJECTIVE: Evaluate whether preemptive pregabalin use compared with placebo decreases pain perception in patients undergoing cardiac surgery in the first 24 hours and 2 months after hospital discharge; evaluate analgesic consumption in the immediate postoperative period; evaluate differences in blood gas parameters between groups; evaluate anesthetic recovery by QoR-40; assess incidence of serious adverse events (reintubation and mental confusion); incidence of delirium through the CAM-ICU questionnaire; assess adverse drug events (nausea, vomiting, pharmacodermia, allergic reactions). METHOD: Randomized, triple-blind, placebo-controlled clinical trial. EXPECTED RESULTS: Postoperative pain control with a drug that could cause fewer side effects, may lead to faster clinical improvement, fewer medications and fewer procedures, and lower healthcare costs with a decrease in intensive care unit (ICU) stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo median sternotomy due to the need for cardiac surgery (valvular or myocardial revascularization);
* Patients between 18 and 70 years old;
* Patients able to swallow tablets and agree to participate in this clinical trial.

Exclusion Criteria:

* Patients with chronic renal failure with creatinine clearance less than or equal to 30 mL/min;
* Patients with known hypersensitivity to pregabalin;
* Hemodynamically unstable patients using vasoactive drugs the day before surgery;
* Unconscious and/or sedated patients, or without cognitive discernment to use the visual analog scale;
* Patients previously submitted to sternotomy; emergency surgery;
* Patients with neurological diseases; anticonvulsant drug users.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception in visual analog scale (0 means no pain and 10 is the most severe pain) at 72 hour post operative | 72 hours post operative
Analgesic opioids consumption at 72 hours post operative | 72 hours post operative

SECONDARY OUTCOMES:
Pain perception in visual analog scale (0 means no pain and 10 is the most severe pain) and analgesic opioids consumption at month 2 post operative | Month 2 post operative
Partial pressure of oxygen in millimeter of mercury (mmHg) | 03 hours, 06 hours, 12 hours and 24 hours post operative
Partial pressure of carbon dioxide in millimeter of mercury (mmHg) | 03 hours, 06 hours, 12 hours and 24 hours post operative
Arterial blood potential of hydrogen (pH) | 03 hours, 06 hours, 12 hours and 24 hours post operative
Oxygen saturation in percentage (%) | 03 hours, 06 hours, 12 hours and 24 hours post operative
Anesthetic recovery by Quality of Recovery 40-item questionnaire (QoR-40 - 40 items questionnaire each item ranging from 1 to 5 being 1 very poor and 5 excellent) | 24 hour post operative
Incidence of serious adverse events (reintubation, infection, bleeding, AKI) | 72 hour post operative
Incidence of delirium by Confusion Assessed Method fo the Intensive Care Unity (CAM-ICU) | 24 hour post operative
Number of participants with treatment-related adverse drug events (nausea, vomiting, pharmacodermia, allergic reactions) assessed by Common Terminology Criteria for Adverse Events (CTCAE v5.0) | 72 hour post operative

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Antonio M Cesar, PhD, Study Director — InCor Heart Institute; Bruno R Barbosa, MD, Principal Investigator — InCor Heart Institute; André T Araújo, PhD, Principal Investigator — UFPB Paraíba Federal University
Locations (2):
- Brazil (2):
  - Hospital João XXIII, Campina Grande, Paraíba
  - Clínica Dom Rodrigo, João Pessoa, Paraíba

IPD SHARING:
Plan to Share IPD: No